CLINICAL TRIAL: NCT06905145
Title: Molecular-Based Selection of Patients with Head and Neck Squamous Cell Carcinoma: Biomarker Analysis
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: MATEs
Record Dates: First submitted 2025-03-18; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Locally Advanced Stage
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group A: Patients undergoing surgery followed by chemo-radiotherapy
  Interventions: Other: Biomarkers evaluation
- Group B: Patients undergoing exclusive chemo-radiotherapy with CDDP, CBDCA, or Cetuximab
  Interventions: Other: Biomarkers evaluation

INTERVENTIONS:
Other: Biomarkers evaluation — Evaluate the prognostic role of the markers TP53, P16, Cyclin D1, EGFR, Akt, PDL-1, ERCC1 examined on biopsy samples.

SUMMARY:
This is an observational, prospective study enrolling patients who meet the inclusion criteria and provide consent for the use of biopsy samples collected as part of standard clinical practice. The analysis will focus on the following biomarkers: TP53, P16, Cyclin D1, EGFR, Akt, PDL-1, and ERCC1.

These biomarkers will be examined in both observation groups.

DETAILED DESCRIPTION:
The primary objective of this project is to evaluate the prognostic role of the biomarker P53, as numerous studies suggest its association with poor prognosis. This analysis will be particularly relevant for p16-positive (HPV-related) patients, who are currently considered a good prognosis category. The study aims to determine whether cases with overexpression of both p16 and P53 deviate from this assumption.

A secondary objective is to validate a molecular signature in clinical practice, composed of multiple biomarkers, to assess whether specific combinations can predict treatment response.

The biomarkers TP53, P16, Cyclin D1, EGFR, Akt, PDL-1, and ERCC1 will be analyzed on biopsy samples from patients with newly diagnosed, locally advanced squamous cell carcinoma of the head and neck.

The study population consists of patients with locally advanced Head and Neck Squamous Cell Carcinoma who have an available biopsy sample collected as part of standard clinical practice. The groups will be classified based on the treatment received:

* Group A: Patients undergoing surgery followed by chemoradiotherapy.
* Group B: Patients receiving exclusive chemoradiotherapy with CDDP, CBDCA, or Cetuximab.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged > 18 years
2. Written informed consent approved by the competent Independent Ethics Committee
3. Histopathological diagnosis of squamous cell carcinoma of the head and neck region originating from one of the following organs or structures: Oral cavity, oropharynx, larynx, hypopharynx
4. Locally advanced stage: from T1N1M0 to T4N3M0
5. Availability of a tissue sample from a biopsy performed according to clinical practice guidelines.

Exclusion Criteria:

1. Recurrent/metastatic disease
2. Presence of a synchronous second tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients with locally advanced Head and Neck Squamous Cell Carcinoma who will have a biopsy sample obtained according to clinical practice. These groups will be divided based on the treatment received:
  * **Group A**: Patients undergoing surgery followed by chemo-radiotherapy
  * **Group B**: Patients undergoing exclusive chemo-radiotherapy with CDDP, CBDCA, or Cetuximab
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of P53 Expression in Tumor Tissue in Groups A and B | 84 months

SECONDARY OUTCOMES:
Overall Survival (OS) | 84 monhts
  Describe the Overall Survival (OS) outcomes obtained in both Groups under observation.
Association between Overall Survival (OS) and the expression of biomarkers | 84 monhts
  Define the association between Overall Survival (OS) and the expression of biomarkers (TP53, P16, Cyclin D1, EGFR, Akt, PDL-1, ERCC1) in both Groups under observation.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Perri, MD, Principal Investigator — IRCCS I.N.T. "G. Pascale"
Locations (1):
- Istituto Nazionale Tumori | "Fondazione Pascale", Napoli, Italy